CLINICAL TRIAL: NCT06326060
Title: Investigation of the Safety and Efficacy of Once Weekly NNC0519-0130 in Participants With Overweight or Obesity - a Dose Finding Study
Brief Title: A Research Study Comparing How Well Different Doses of the Medicine NN0519-0130 Help People With Excess Body Weight Lose Weight
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9541-5015; U1111-1291-9210 (Other: World Health Organization (WHO)); jRCT2051230198 (Registry Identifier: JRCT)
Record Dates: First submitted 2024-03-16; First posted 2024-03-22 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- Dosing scheme a: NNC0519-0130 (Experimental): Participants will receive NNC0519-0130 at 1 dose level subcutaneously (s.c.) once-weekly up to 36 weeks.
  Interventions: Drug: NNC0519-0130
- Dosing scheme a: Placebo (Placebo Comparator): Participants will receive NNC0519-0130 matched placebo s.c. once-weekly up to 36 weeks.
  Interventions: Drug: Placebo
- Dosing scheme b: NNC0519-0130 (Experimental): Participants will receive NNC0519-0130 at 2 dose levels s.c. once-weekly up to 36 weeks.
  Interventions: Drug: NNC0519-0130
- Dosing scheme b: Placebo (Placebo Comparator): Participants will receive NNC0519-0130 matched placebo s.c. once-weekly up to 36 weeks.
  Interventions: Drug: Placebo
- Dosing scheme c: NNC0519-0130 (Experimental): Participants will receive NNC0519-0130 at 3 dose levels s.c. once-weekly up to 36 weeks.
  Interventions: Drug: NNC0519-0130
- Dosing scheme c: Placebo (Placebo Comparator): Participants will receive NNC0519-0130 matched placebo s.c. once-weekly up to 36 weeks.
  Interventions: Drug: Placebo
- Dosing scheme d: NNC0519-0130 (Experimental): Participants will receive NNC0519-0130 at 4 dose levels s.c. once-weekly up to 36 weeks.
  Interventions: Drug: NNC0519-0130
- Dosing scheme d: Placebo (Placebo Comparator): Participants will receive NNC0519-0130 matched placebo s.c. once-weekly up to 36 weeks.
  Interventions: Drug: Placebo
- Dosing scheme e: NNC0519-0130 (Experimental): Participants will receive NNC0519-0130 at 5 dose levels s.c. once-weekly up to 36 weeks.
  Interventions: Drug: NNC0519-0130
- Dosing scheme e: Placebo (Placebo Comparator): Participants will receive NNC0519-0130 matched placebo s.c. once-weekly up to 36 weeks.
  Interventions: Drug: Placebo
- Dosing scheme f: NNC0519-0130 (Experimental): Participants will receive NNC0519-0130 at 6 dose levels s.c. once-weekly up to 36 weeks.
  Interventions: Drug: NNC0519-0130
- Dosing scheme f: Placebo (Placebo Comparator): Participants will receive NNC0519-0130 matched placebo s.c. once-weekly up to 36 weeks.
  Interventions: Drug: Placebo
- Dosing scheme g: Tirzepatide (Active Comparator): Participants will receive tirzepatide at 6 dose levels s.c. once weekly up to 36 weeks.
  Interventions: Drug: Tirzepatide

INTERVENTIONS:
Drug: NNC0519-0130 — NNC0519-0130 will be administered subcutaneously.
  Arms: Dosing scheme a: NNC0519-0130; Dosing scheme b: NNC0519-0130; Dosing scheme c: NNC0519-0130; Dosing scheme d: NNC0519-0130; Dosing scheme e: NNC0519-0130; Dosing scheme f: NNC0519-0130
Drug: Placebo — Placebo will be administered subcutaneously.
  Arms: Dosing scheme a: Placebo; Dosing scheme b: Placebo; Dosing scheme c: Placebo; Dosing scheme d: Placebo; Dosing scheme e: Placebo; Dosing scheme f: Placebo
Drug: Tirzepatide — Tirzepatide will be administered subcutaneously.
  Arms: Dosing scheme g: Tirzepatide

SUMMARY:
This study will look at how a new medicine called NNC0519-0130 helps people with excess body weight lose weight. The study will test up to 6 different doses of NNC0519-0130. Participants will take 1-2 injections once a week. The study medicine will be injected under skin with a thin needle in the stomach, thigh, or upper arm. The study will last for about 42 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Female of non-childbearing potential, or male.

  a. For US only: Female of childbearing potential using highly effective non-systemic methods of contraception with low user-dependency at least 2 months prior to screening and willingness to continue using it through-out the study, or male.
* Age 18-75 years (both inclusive) at the time of signing the informed consent.
* History of at least one self-reported unsuccessful dietary effort to lose body weight.
* a) BMI ≥ 27.0 kg/m2 with the presence of at least one weight-related co-morbidity including, but not limited to, hypertension, dyslipidaemia, obstructive sleep apnoea or cardiovascular disease.
* b) BMI ≥ 30.0 kg/m2.

Exclusion Criteria:

* HbA1c greater than equal to 6.5% (48 millimoles per mole (mmol/mol)) as measured by the central laboratory at screening.
* History of type 1 or type 2 diabetes mellitus.
* Treatment with any medication prescribed for the indication of obesity or weight management within 90 days before screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2024-03-18 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Relative change in body weight | From baseline (week 0) to end of treatment (week 36)
  Measured in percentage of body weight.

SECONDARY OUTCOMES:
Change in body weight | From baseline (week 0) to end of treatment (week 36)
  Measured in kilograms (kg)
Achievement of greater than equal to (≥) 5% weight reduction | From baseline (week 0) to end of treatment (week 36)
  Count of participants
Achievement of ≥ 10% weight reduction | From baseline (week 0) to end of treatment (week 36)
  Count of participants
Achievement of ≥ 15% weight reduction | From baseline (week 0) to end of treatment (week 36)
  Count of participants
Achievement of ≥ 20% weight reduction | From baseline (week 0) to end of treatment (week 36)
  Count of participants
Change in body mass index (BMI) | From baseline (week 0) to end of treatment (week 36)
  Measured in Kilogram per meter square (Kg/m^2)
Change in waist circumference | From baseline (week 0) to end of treatment (week 36)
  Measured in centimeter (cm)
Change in glycated hemoglobin (HbA1c) | From baseline (week 0) to end of treatment (week 36)
  Measured in percentage point (%-point)
Change in fasting plasma glucose (FPG) | From baseline (week 0) to end of treatment (week 36)
  Measured in millimoles per liter (mmol/L)
Change in systolic blood pressure (SBP) | From baseline (week 0) to end of treatment (week 36)
  Measured in milliters of mercury (mmHg)
Change in high sensitivity C-Reactive protein (hsCRP) | From baseline (week 0) to end of treatment (week 36)
  Ratio to baseline
Change in total cholesterol | From baseline (week 0) to end of treatment (week 36)
  Ratio to baseline
Change in high-density lipoprotein (HDL) cholesterol | From baseline (week 0) to end of treatment (week 36)
  Ratio to baseline
Change in low-density lipoprotein (LDL) cholesterol | From baseline (week 0) to end of treatment (week 36)
  Ratio to baseline
Change in triglycerides | From baseline (week 0) to end of treatment (week 36)
  Ratio to baseline
Change in Impact of Weight on Quality of Life-Lite Clinical Trials (IWQOL-Lite-CT) Physical composite score | From baseline (week 0) to end of treatment (week 36)
  IWQOL-Lite-CT measures weight-related physical and psychosocial functioning. The measure consists of 20 items yielding 3 composite scores, and 1 total score. Higher scores indicate better levels of functioning. Total score range is 0-100. Composite score ranges are: physical composite (0-100), psychosocial composite (0-100), and physical function composite (0-100).
Change in IWQOL-Lite-CT Psychosocial composite score | From baseline (week 0) to end of treatment (week 36)
  IWQOL-Lite-CT measures weight-related physical and psychosocial functioning. The measure consists of 20 items yielding 3 composite scores, and 1 total score. Higher scores indicate better levels of functioning. Total score range is 0-100. Composite score ranges are: physical composite (0-100), psychosocial composite (0-100), and physical function composite (0-100).
Change in IWQOL-Lite-CT Physical Function score | From baseline (week 0) to end of treatment (week 36)
  IWQOL-Lite-CT measures weight-related physical and psychosocial functioning. The measure consists of 20 items yielding 3 composite scores, and 1 total score. Higher scores indicate better levels of functioning. Total score range is 0-100. Composite score ranges are: physical composite (0-100), psychosocial composite (0-100), and physical function composite (0-100).
Change in IWQOL-Lite-CT Total score | From baseline (week 0) to end of treatment (week 36)
  IWQOL-Lite-CT measures weight-related physical and psychosocial functioning. The measure consists of 20 items yielding 3 composite scores, and 1 total score. Higher scores indicate better levels of functioning. Total score range is 0-100. Composite score ranges are: physical composite (0-100), psychosocial composite (0-100), and physical function composite (0-100).
Number of adverse events | From baseline (week 0) to end of treatment (week 40)
  Count of events

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (51):
- United States (39):
  - Centricity Research-Arizona, Mesa, Arizona
  - Arkansas Clinical Research, Little Rock, Arkansas
  - Unity Health-Searcy Medical Center, Searcy, Arkansas
  - FDRC, Costa Mesa, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Univ of Colorado at Denver, Aurora, Colorado
  - Nature Coast Clinical Research, Crystal River, Florida
  - Northeast Research Institute, Fleming Island, Florida
  - Jacksonville Ctr For Clin Res, Jacksonville, Florida
  - Cedar-Crosse Research Center, Chicago, Illinois
  - Midwest Inst For Clin Res, Indianapolis, Indiana
  - Velocity Clin. Res Valparaiso, Valparaiso, Indiana
  - L-MARC Research Center, Louisville, Kentucky
  - Centennial Medical Group, Columbia, Maryland
  - StudyMetrix Research LLC, City of Saint Peters, Missouri
  - NYU Bariatric Surgical Ctr, New York, New York
  - Medication Mgmnt, LLC_Grnsboro, Greensboro, North Carolina
  - PharmQuest Life Sciences LLC, Greensboro, North Carolina
  - Physicians East Endocrinology, Greenville, North Carolina
  - Piedmont Healthcare, Statesville, North Carolina
  - Accellacare, Wilmington, North Carolina
  - Remington Davis Inc, Columbus, Ohio
  - Family Practice Center of Wadsworth Inc., Wadsworth, Ohio
  - Lynn Institute of Norman, Norman, Oklahoma
  - The University of Penn Center, Philadelphia, Pennsylvania
  - Preferred Primary Care Physicians_Pittsburgh, Pittsburgh, Pennsylvania
  - Velocity Clin Res Providence, East Greenwich, Rhode Island
  - Medical University Of South Carolina, Charleston, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Holston Medical Group Pc, Bristol, Tennessee
  - Baylr Sctt White Rs Inst, Endo, Dallas, Texas
  - Velocity Clinical Res-Dallas, Dallas, Texas
  - North Texas Endocrine Center, Dallas, Texas
  - UT Southwestern Medical Center - Lingvay, Dallas, Texas
  - DCOL Ctr for Clin Res, Longview, Texas
  - Washington Cntr Weight Mgmt, Arlington, Virginia
  - Health Res of Hampton Roads, Newport News, Virginia
  - TPMG Clinical Research, Newport News, Virginia
  - National Clin Res Inc., Richmond, Virginia
- Australia (10):
  - Paratus Clinical, Blacktown, New South Wales
  - Northern Beaches Clinical Research, Brookvale, New South Wales
  - Momentum Clinical Research Darlinghurst, Darlinghurst, New South Wales
  - Novatrials, Kotara, New South Wales
  - Paratus Clinical, Herston, Queensland
  - University of Sunshine Coast, Sippy Downs, Queensland
  - CMAX Clinical Research, Norwood, South Australia
  - Emeritus Research Melbourne, Camberwell, Victoria
  - Austin Health, Metabolic Disorders Centre, Heidelberg Heights, Victoria
  - Linear Clinical Research, Nedlands, Western Australia
- Japan (2):
  - OCROM Clinic, Suita-shi, Osaka
  - ToCROM Clinic, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com